CLINICAL TRIAL: NCT03737916
Title: To Evaluate the Effect of Perineural Dextrose Injection in Patients With Ulnar Neuropathy at the Elbow and to Compare the Control Group
Brief Title: The Effect of Perineural Dextrose Injection in Patients With Ulnar Neuropathy at the Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Basak Mansiz-Kaplan, Department of Physical Medicine and Rehabilitation (the principal investigator), Ankara Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E171616
Record Dates: First submitted 2018-11-06; First posted 2018-11-13 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Ulnar Neuropathies
MeSH Terms: conditions — Ulnar Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dextrose group (Experimental): Procedure: Ultrasound-guided perineural injection with 5% dextrose. Ultrasound-guided perineural injection with 5% Dextrose (1cc) to ulnar nerve into the elbow, 2 and 4 cm before and after the elbow (total 5 cc).
  Drug: 5% Dextrose 5% Dextrose could decrease the release of CGRP (Calcitonin Gene Related Peptide) and substance P to reduce the nerve inflammation
  Interventions: Other: 5 cc 5% Dextrose solution
- control group (Placebo Comparator): Procedure: Perineural injection with normal saline Ultrasound-guided perineural injection with normal saline (1cc) to ulnar nerve into the elbow, 2 and 4 cm before and after the elbow (total 5 cc).
  Drug: Normal Saline Normal saline is safe for perineural injection.
  Interventions: Other: 5 cc salin

INTERVENTIONS:
Other: 5 cc 5% Dextrose solution — Ultrasound-guided perineural injection with 5% Dextrose (1cc) to ulnar nerve into the elbow, 2 and 4 cm before and after the elbow (total 5 cc).
  Arms: dextrose group
Other: 5 cc salin — Ultrasound-guided perineural injection with salin (1cc) to ulnar nerve into the elbow, 2 and 4 cm before and after the elbow (total 5 cc).
  Arms: control group

SUMMARY:
Ulnar neuropathy at the elbow (UNE) is the second most common neuropathy and occurs after recurrent or elongated elbow flexion. Diagnosis of UNE depends on clinical symptoms, physical examination, and electrophysiological findings. Imaging methods such as ultrasonography (USG) and magnetic resonance imaging show cross-sectional area and echogenicity of ulnar nerve and give information about to surrounding structures around the ulnar nerve. In mild and moderate cases, conservative treatments are administered up to 6 months, who do not benefit from conservative treatment are referred to surgery. There are not many options for conservative treatment. Activity modification, nerve gliding exercises and night splints are conservative treatment methods. Steroid injection is no longer recommended. Perineural dextrose injection is applied in tendinopathies and entrapment neuropathies (especially carpal tunnel syndrome). In the literature, there is no study showing effect of perineural dextrose injection in patients with UNE. The investigators design a randomized, double-blind, controlled trail to evaluate the effect after ultrasound-guided perineural injection with 5% dextrose in patients with UNE.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients of clinically diagnosed with UNE were randomized into intervention and control group. Participants in intervention group received one-session ultrasound-guided perineural injection with 5% dextrose and control group received one-session ultrasound-guided perineural injection with normal saline. No additional treatment after injection through the study period. The primary outcome is visual analog scale (VAS) and secondary outcomes include Quick-DASH (Disabilities of Arm, Shoulder and Hand), cross-sectional area (CSA) of the ulnar nerve, motor nerve conduction velocity and distal latency of the ulnar nerve. The evaluation was performed pretreatment as well as on the 2nd week, 1st and 3rd month after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 year-old.
* Neuropathic pain on the ulnar nerve distribution area for at least 1 months
* Diagnosis was confirmed using an electrophysiological studies and ultrasonography

Exclusion Criteria:

* History of trauma to the upper extremity
* Central or peripheral neurologic disease
* Electromyography (EMG)-proven carpal tunnel syndrome, radiculopathy or any other neuropathy
* Pregnancy or any systemic disease that might cause swelling on nerves (e.g., diabetes -mellitus, renal failure, and thyroid disease)
* USG-detected bifid or trifid median nerve, persistent median artery, or space-occupying lesions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 2nd week, 1st and 3rd months after treatment: VAS | Time Frame: Pre-treatment, 2nd week, 1st and 3rd months after treatment
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment. Recorded on a visual analogue scale (VAS), scores range from 0 to 100 mm, with higher scores indicating worse pain.

SECONDARY OUTCOMES:
Change from baseline in activity and functional status on 2nd week, 1st and 3rd months after treatment. | Pre-treatment, 2nd week, 1st and 3rd months after treatment
  Using the Quick-DASH to measure the activity and functional status before treatment and multiple time frame after treatment. The Quick-DASH is a shortened version of the DASH Outcome Measure. Instead of 30 items, the QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. The higher scores indicate worse functional status.
Change from baseline in cross-sectional area of the ulnar nerve on 1st and 3th months after treatment. | Pre-treatment, 2nd week, 1st and 3rd months after treatment treatment
  Using the musculoskeletal ultrasonography to measure the cross-sectional area of the ulnar nerve.
Change from baseline in motor nerve conduction velocity of the ulnar nerve | Pre-treatment, 1st and 3rd months after treatment treatment
  Using Electromyography to measure the motor nerve conduction velocity (m/sn) of the ulnar nerve

CONTACTS AND LOCATIONS:
Overall Officials: Basak Mansiz-Kaplan, M.D., Principal Investigator — Department of Physical Medicine and Rehabilitation
Locations (1):
- Basak Mansiz-Kaplan, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Mansiz-Kaplan B, Nacir B, Pervane-Vural S, Tosun-Meric O, Duyur-Cakit B, Genc H. Effect of Perineural Dextrose Injection on Ulnar Neuropathy at the Elbow: A Randomized, Controlled, Double-Blind Study. Arch Phys Med Rehabil. 2022 Nov;103(11):2085-2091. doi: 10.1016/j.apmr.2022.04.013. Epub 2022 Jun 9. PMID 35690093